CLINICAL TRIAL: NCT06439277
Title: Efficacy and Safety of Tirzepatide Once Weekly Versus Placebo for the Treatment of Obesity and Weight-Related Comorbidities in Adolescents: A Randomized, Double-Blind, Placebo- Controlled Trial (SURMOUNT-ADOLESCENTS-2)
Brief Title: A Study of Tirzepatide in Adolescents With Obesity and Weight-Related Comorbidities (SURMOUNT-ADOLESCENTS-2)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18832; I8F-MC-GPIX (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-05-28; First posted 2024-06-03 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Obesity; Weight Gain
MeSH Terms: conditions — Obesity; Weight Gain | interventions — Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tirzepatide (Experimental): Participants will receive tirzepatide subcutaneously (SC).
  Interventions: Drug: Tirzepatide
- Placebo (Placebo Comparator): Participants will receive placebo SC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176
  Arms: Tirzepatide
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The goal of the study is to assess how tirzepatide impacts bodyweight and cardiovascular risk factors when used in conjunction with healthy nutrition and physical activity in adolescents with obesity and multiple weight related comorbidities. The study will last approximately 76 weeks and may include up to 23 visits.

Participants who have completed the primary 72-week GPIX study and have been off treatment for no more than 12 weeks (including the 4-week safety follow-up period), will have the opportunity to receive an additional 156 weeks of treatment with tirzepatide as well as continuing the lifestyle intervention.

DETAILED DESCRIPTION:
The main purpose of this study is to evaluate the safety and efficacy of tirzepatide in adolescents that have obesity with multiple weight related comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* Have body mass index (BMI) equal to or above the 95th percentile for age and sex (on age and gender-specific growth chart for diagnosis of obesity) with at least 2 of the following predefined weight-related comorbidities: hypertension, prediabetes and hypertriglyceridemia.
* Have history of at least 1 self-reported unsuccessful dietary effort to lose weight.
* Are capable of giving signed informed consent by a legal representative or assent by a study participant (when applicable).

Exclusion Criteria:

* Have undergone or plan to undergo a weight reduction procedure during the study, such as, but not limited to

  * gastric bypass
  * sleeve gastrectomy
  * restrictive bariatric surgery, such as Lap-Band gastric banding, or
  * any other procedure intended to result in weight reduction.
* Have a self-reported, or by parent or legal guardian where applicable, decrease in body weight greater than 5 kg (11 lbs) within 90 days before screening irrespective of medical records
* Have type 1 diabetes or history of ketoacidosis, or hyperosmolar state
* Have type 2 diabetes or have a HbA1c > 6.4% at screening
* Have a history of chronic or acute pancreatitis
* Have a family or personal history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome type 2

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Percent Change from Baseline in Body Mass Index (BMI) | Baseline, Week 72
A Composite Endpoint of Normalization or Clinically Significant Improvement in At Least 2 Predefined Weight-Related Comorbidities Present at Screening Without Development of New Predefined Comorbidity or Worsening of Existing Predefined Comorbidity | Baseline, Week 72

SECONDARY OUTCOMES:
Percentage of Participants Who Achieve BMI Reduction of ≥ 5% | Week 72
Percentage of Participants Who Achieve BMI Reduction of ≥ 10% | Week 72
Percentage of Participants Who Achieve BMI Reduction of ≥ 15% | Week 72
Percentage of Participants Who Achieve BMI Reduction of ≥ 20% | Week 72
Change from Baseline in Hemoglobin A1c (HbA1c) | Baseline, Week 72
Percent Change from Baseline in Triglycerides | Baseline, Week 72
Change from Baseline in Systolic Blood Pressure (SBP) | Baseline, Week 72
Change from Baseline in Peripheral Apnea-Hypopnea Index (pAHI) | Baseline, Week 72
Percent Change from Baseline in Total Body Fat Mass as Determined by Dual energy X-ray Absorptiometry (DXA) | Baseline, Week 72
Change from Baseline in Diastolic Blood Pressure (DBP) | Baseline, Week 72
Percent Change from Baseline in Body Weight | Baseline, Week 72
Change from Baseline in Waist Circumference | Baseline, Week 72

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (75):
- United States (15):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Sutter Valley Medical Foundation (SVMF) Pediatric Endocrinology, Sacramento, California
  - Nemours Children's Health - Delaware, Wilmington, Delaware
  - CenExel iResearch, LLC, Decatur, Georgia
  - Medical Research Partners, Ammon, Idaho
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Indiana University Health University Hospital, Indianapolis, Indiana
  - UBMD Pediatrics, Buffalo, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Epic Medical Research - DeSoto, DeSoto, Texas
  - Valley Institute of Research - Fort Worth, Fort Worth, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - Texas Valley Clinical Research, Weslaco, Texas
  - Alliance for Multispecialty Research, LLC, Layton, Utah
- Argentina (6):
  - Investigaciones Medicas Imoba Srl, Buenos Aires
  - Centro de Investigaciones Metabólicas (CINME), Buenos Aires
  - Centro Medico Dra. Laura Maffei- Investigacion Clinica Aplicada, Buenos Aires
  - Fundación Respirar, Buenos Aires
  - DIM Clínica Privada, Ramos Mejía
  - Centro de Investigaciones Médicas Tucuman, SAN M. de Tucuman
- Australia (6):
  - Nightingale Research, Adelaide
  - Cornerstone Dermatology, Coorparoo
  - Hunter Medical Research Institute, Newcastle
  - Perth Children's Hospital, Perth
  - University of Sydney - Charles Perkins Centre, Sydney
  - The Children's Hospital at Westmead, Westmead
- Canada (4):
  - Alberta Children's Hospital, Calgary
  - Winterberry Research Inc., Hamilton
  - Premier Clinical Trial Network, Hamilton
  - Bluewater Clinical Research Group Inc., Sarnia
- France (7):
  - Centre Hospitalier Universitaire d'Angers, Angers
  - Hospices Civils de Lyon - Hopital Louis Pradel, Bron
  - Hôpital Jeanne de Flandre, Lille
  - Assistance Publique Hôpitaux de Marseille - Hôpital de la Timone, Marseille
  - Hôpital Armand Trousseau, Paris
  - Assistance Publique - Hopitaux de Paris (AP-HP) - Hopital Robert Debre - Centre Hospitalo Universitaire (C -T, Paris
  - CHU de Toulouse - Hôpital des Enfants, Toulouse
- Germany (3):
  - Universitaetsklinikum Koeln, Cologne
  - Universitätsklinikum Leipzig, Leipzig
  - Universitaetsklinikum Ulm, Ulm
- Israel (9):
  - Emek Medical Center, Afula
  - Yitzhak Shamir Medical Center, Beer Yaacov
  - Soroka Medical Center, Beersheba
  - Rambam Health Care Campus, Haifa
  - Carmel Hospital, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Schneider Children's Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
- Mexico (5):
  - Centro de Atención e Investigación Clínica, Aguascalientes
  - Centro de Investigacion Medica de Occidente, S.C., Guadalajara
  - Christus - Latam Hub Center of Excellence and Innovation S.C., Monterrey
  - Clínica García Flores SC, Monterrey
  - Consultorio Médico de Endocrinología y Pediatría, Puebla City
- University Pediatric Hospital, San Juan, Puerto Rico
- Spain (6):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Infantil Universitario Niño Jesús, Madrid
  - H.R.U Málaga - Hospital General, Málaga
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
- Taiwan (4):
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District
- United Kingdom (9):
  - Addenbrooke's Hospital, Cambridge
  - Royal Hospital for Children, Glagow
  - Leeds General Infirmary, Leeds
  - Leicester Royal Infirmary, Leicester
  - Alder Hey Children's Hospital, Liverpool
  - Paediatric and Adolescent OutpatientsElizabeth Garrett Anderson WingUniversity College Hospital, London
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Sheffield Children's Hospital, Sheffield
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of Tirzepatide in Adolescents With Obesity and Weight-Related Comorbidities (SURMOUNT-ADOLESCENTS-2) — https://trials.lilly.com/en-US/trial/494896